CLINICAL TRIAL: NCT05521971
Title: The Impact of a Pharmacist Intervention on Post-discharge Hypnotic Drug Discontinuation in Geriatric Inpatients: a Before-after Study
Brief Title: The Impact of a Pharmacist Intervention on Post-discharge Hypnotic Drug Discontinuation in Geriatric Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: S59134
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hypnotic Withdrawal
Keywords: deprescribing; tapering; adverse events; hypnotics; benzodiazepines; z-drugs; geriatrics

STUDY DESIGN:
Intervention Model Description: before-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Before group (Other): In the usual care cohort, there was no systematic clinical pharmacist involvement regarding deprescribing of hypnotics.
  Interventions: Other: Usual care group
- After group (Experimental): In the intervention cohort a pharmacist-led intervention was implemented comprising the four following components: 1) education of health care personnel; 2) access to standardized discontinuation regimens; 3) patient education; 4) support of transitional care.
  Interventions: Other: multifaceted pharmacist-led intervention

INTERVENTIONS:
Other: multifaceted pharmacist-led intervention — * Educational sessions were provided to the physicians and nursing staff.
  * Discontinuation regimens were developed. Prescribers were free to choose whether or not to actually use them. The regimens were derived from the regimen used by Petrovic et al. and encouraged a switch from any benzodiazepine to lorazepam 1 mg OD for one week followed by drug stop. Z-drugs were switched to zolpidem 5 mg OD for one week followed by drug stop. If deemed necessary, a pro re nata regimen of lorazepam 1 mg or zolpidem 5 mg for one additional week was prescribed respectively. The discontinuation regimens were incorporated into the hospital's electronic prescribing system. Furthermore, a clinical decision support system provided additional support.
  * Patient education sessions were provided upon enrolment and at discharge. Specific patient leaflets were used to facilitate patient education.
  * The patient's primary care physician and, if applicable, the nursing home were informed by phone.
  Arms: After group
Other: Usual care group — all patients received comprehensive geriatric care without any systematic clinical pharmacist involvement regarding deprescribing of hypnotics. Treating physicians were not actively informed on the patient's participation in this particular study.
  Arms: Before group

SUMMARY:
This study investigated whether a multifaceted approach was associated with hypnotic drug discontinuation at one month after discharge

DETAILED DESCRIPTION:
Chronic use of hypnotic agents is prevalent in older adults, who as a result are at increased risk for certain adverse events, such as day-time drowsiness and falls. Multiple strategies to discontinue hypnotics have been tested in geriatric patients, but evidence remains scarce. Hence, we aimed to investigate a multicomponent intervention to reduce hypnotic drug use in geriatric inpatients.

A before-after study was performed on the acute geriatric wards of a teaching hospital. The before cohort received usual care while intervention patients were exposed to a pharmacist-led deprescribing intervention, comprising education of health care personnel, access to standardized discontinuation regimens, active patient involvement and support of transitional care. The primary outcome was hypnotic drug discontinuation at one month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 75 years
* Admitted to an acute geriatric ward of UZ Leuven
* Documented chronic use of a hypnotic drug (hypnotics were defined as benzodiazepines and Z-drugs and chronic hypnotic drug use was defined as hypnotic use for at least five days a week during a minimum of four consecutive weeks.
* Indication: insomnia, anxiety or an undefined reason

Exclusion Criteria:

* Concomitant use of multiple benzodiazepines and/or Z-drugs
* Discontinuation of the hypnotic drug prior to enrollment
* Estimated discharge from the hospital within 72 hours of admission
* No command of the Dutch language
* Severe psychiatric or neurological disease (e.g. bipolar disorder, epilepsy or dystonia) or a severe acute medication condition in the opinion of the treating physician
* End-of-life care.

Study participants who died during their hospital stay were excluded from the analysis as their medication at discharge could not be evaluated. In case of any readmission, only the first admission was included in the analysis.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 173 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Hypnotic drug discontinuation at one month after discharge | 1 month after discharge
  Difference in hypnotic discontinuation rate between before and after group

SECONDARY OUTCOMES:
Hypnotic drug use | 1 and 2 weeks after enrollment and at discharge (the end of the hospital stay, on average 12 days after admission)
  Description of type and dose of hypnotic drug use
Restart of hypnotics during hospital stay | From enrollment until discharge (the end of the hospital stay, on average 12 days after admission)
  The emergency use of hypnotics after any discontinuation attempt during hospital stay.
Safety - incidence of delirium occurence during hospital stay | From enrollment until discharge (the end of the hospital stay, on average 12 days after admission)
  During hospital stay the incidence of physician-identified delirium was assessed together with emergency use of antipsychotics
Sleep quality | Upon inclusion, fourteen days after enrollment and one month after discharge
  Sleep quality was determined during a patient interview using the Pittsburgh Sleep Quality Index (PSQI). The PSQI concerns a validated questionnaire where a higher score signifies a worse sleep quality; a total score of 5 or more indicates poor sleep quality
Fall risk | 1 month after discharge
  The occurrence of falls
Determinants for post-discharge hypnotic discontinuation | 1 month after discharge
  Factors associated with hypnotic discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jos Tournoy, Prof, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No
Only upon reasonable request

REFERENCES:
- [Background] Petrovic M, Pevernagie D, Mariman A, Van Maele G, Afschrift M. Fast withdrawal from benzodiazepines in geriatric inpatients: a randomised double-blind, placebo-controlled trial. Eur J Clin Pharmacol. 2002 Jan;57(11):759-64. doi: 10.1007/s00228-001-0387-4. PMID 11868796
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Derived] Van der Linden L, Hias J, Liesenborghs A, Walgraeve K, Van Brantegem P, Hellemans L, Milisen K, Tournoy J. The impact of a pharmacist intervention on post-discharge hypnotic drug discontinuation in geriatric inpatients: a before-after study. BMC Geriatr. 2023 Jul 4;23(1):407. doi: 10.1186/s12877-023-04139-y. PMID 37400758